CLINICAL TRIAL: NCT06978166
Title: Evaluating and Optimizing Just-In-Time Adaptive Interventions (JITAIs) in a Digital Mental Health Intervention (Wysa for Chronic Pain) for Middle-Aged and Older Adults With Chronic Pain
Brief Title: Just-In-Time Adaptive Interventions (JITAIs) in a Digital Mental Health Intervention for Middle-Aged and Older Adults With Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Duke University (Other); Wysa (Industry)
Responsible Party: Principal Investigator, Abby Cheng, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00085039; R01MH131989 (NIH)
Record Dates: First submitted 2025-05-05; First posted 2025-05-18 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Depression, Anxiety
Keywords: JITAI; Digital mental health intervention; Older adults; Middle-aged adults; App; Smartphone; Chronic pain; Depression; Anxiety; Chatbot
MeSH Terms: conditions — Chronic Pain; Depression; Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wysa for Chronic Pain + JITAIs (Experimental): Participants assigned to the experimental arm will receive access to the Wysa for Chronic Pain app, and the novel JITAIs that are being tested in this study will be incorporated into the app experience.
  In an initial 4-week pilot trial, participants in this arm will receive the JITAIs every time the decision rule (i.e., "trigger criteria") is satisfied for that respective JITAI. In subsequent 12-week micro-randomized trials, every time the decision rule for a JITAI is satisfied, participants in this arm will be randomized to receive (versus not receive) the respective JITAI.
  Interventions: Other: Just-In-Time Adaptive Interventions (JITAIs); Behavioral: Wysa for Chronic Pain
- Wysa for Chronic Pain without JITAIs (Active Comparator): Participants assigned to the control arm will receive access to the Wysa for Chronic Pain app, but the novel JITAIs that are being tested in this study will not be incorporated into the app experience.
  Interventions: Behavioral: Wysa for Chronic Pain

INTERVENTIONS:
Other: Just-In-Time Adaptive Interventions (JITAIs) — JITAIs are digital interventions that aim to deliver support to a user when the person is most in need and receptive to the intervention. In this study, multiple JITAIs will be tested and refined through completion of an iterative series of randomized trials that are interspersed with qualitative participant interviews. The purpose of each JITAI under investigation is to improve engagement with the Wysa for Chronic Pain app.
  Arms: Wysa for Chronic Pain + JITAIs
Behavioral: Wysa for Chronic Pain — Wysa for Chronic Pain is an app-based digital mental health intervention that uses a behavioral activation framework and encourages users to work toward pain acceptance. The intervention also includes cognitive behavioral therapy, mindfulness, and sleep tools.

SUMMARY:
The purpose of this research study is to refine customized in-app notifications in order to optimize users' experience with a mobile app called Wysa for Chronic Pain. This app is designed to support people who have chronic pain and who also experience symptoms of depression and/or anxiety. This version of the app is not currently available to the public. Eligible participants will be asked to download and use the Wysa for Chronic Pain study app for several weeks, and to use it as they normally would if they were not part of a research study. At the beginning and end of the study period, participants will be asked to complete brief surveys about their mood, pain, physical function, and sleep. Additionally, a few participants will be asked to share their experience with the study app at the end of the research study in a casual interview using a secure audio/video recorded call. Participating in the interview portion is optional.

ELIGIBILITY:
Inclusion Criteria:

* 45 years or older
* At least moderately severe depression and/or anxiety symptoms (Patient Health Questionnaire-9 (PHQ-9) and/or Generalized Anxiety Disorder-7 (GAD-7) score ≥ 10)
* Chronic pain (i.e., pain on most days or every day in the past three months)

Exclusion Criteria:

* Frequent active suicidal ideation
* No access to a mobile device
* Not living in the United States

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Engagement | Each JITAI has a different target engagement time interval. e.g., varying from 24 hours to 7 days.
  The primary outcome for each JITAI is the between-group difference in engagement with Wysa for Chronic Pain during the JITAI's target engagement time interval. Engagement is operationalized as interaction(s) with the digital mental health intervention and is automatically captured throughout the study by the intervention's technical infrastructure. It is not self-reported.

OTHER OUTCOMES:
Patient Health Questionnaire Anxiety-Depression Scale (PHQ-ADS) | Baseline, Week 4, Week 8 (Not in pilot trial), Week 12 (Not in pilot trial)
  The PHQ-ADS will be collected as the distal clinical outcome. It is a16-item self-reported measure that is used to assess depression and anxiety symptoms. Scores range from 0 to 48, and higher scores indicate more distress.

CONTACTS AND LOCATIONS:
Overall Officials: Abby L. Cheng, MD, MPHS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data will be shared through the NIMH Data Archive (NDA). Access to the dataset will be managed by the NDA.

REFERENCES:
- [Derived] Cheng AL, Abraham J, Hartz SM, Laber EB, Miller JP. Evaluating and Optimizing Just-in-Time Adaptive Interventions in a Digital Mental Health Intervention (Wysa for Chronic Pain) for Middle-Aged and Older Adults With Chronic Pain: Protocol for a Series of Randomized Trials. JMIR Res Protoc. 2025 Sep 17;14:e77532. doi: 10.2196/77532. PMID 40961490